CLINICAL TRIAL: NCT02332720
Title: A Phase II, Randomized, Open-Label Clinical Trial to Study the Efficacy and Safety of the Combination Regimen of MK-5172 and MK-3682 With Either MK-8742 or MK-8408 in Subjects With Chronic HCV GT3, GT4, GT5, and GT6 Infection
Brief Title: Efficacy and Safety of Grazoprevir (MK-5172) and Uprifosbuvir (MK-3682) With Elbasvir (MK-8742) or Ruzasvir (MK-8408) for Chronic Hepatitis C Virus (HCV) Genotype (GT) 3, GT4, GT5, and GT6 Infection (MK-3682-012)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3682-012; 2014-003347-35 (EudraCT Number)
Record Dates: First submitted 2015-01-06; First posted 2015-01-07 (Estimated); Results first posted 2018-07-02 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — grazoprevir; uprifosbuvir; elbasvir; ruzasvir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (22):
- A1: GT3 NC TN Grazoprevir+Uprifosbuvir+Elbasvir (8 weeks) (Experimental): In Part A, HCV GT3-infected NC TN participants will take grazoprevir (100 mg) + uprifosbuvir (300 mg) + elbasvir (50 mg) q.d. by mouth for 8 weeks. Part A participants who relapsed following completion of therapy were offered the option of retreatment with 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d. and RBV (weight-based dosing) b.i.d. by mouth for 16 weeks during Part C.
  Interventions: Drug: Grazoprevir; Drug: Uprifosbuvir; Drug: Elbasvir; Drug: MK-3682B; Drug: Ribavirin (RBV)
- A2: GT3 NC TN Grazoprevir+Uprifosbuvir+Ruzasvir (8 weeks) (Experimental): In Part A, HCV GT3-infected NC TN participants will take grazoprevir (100 mg) + uprifosbuvir (300 mg) + ruzasvir (60 mg) q.d. by mouth for 8 weeks. Part A participants who relapsed following completion of therapy were offered the option of retreatment with 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d. and RBV (weight-based dosing) b.i.d. by mouth for 16 weeks during Part C.
  Interventions: Drug: Grazoprevir; Drug: Uprifosbuvir; Drug: Ruzasvir; Drug: MK-3682B; Drug: Ribavirin (RBV)
- A3: GT3 NC TN Grazoprevir+Uprifosbuvir+Elbasvir (8 weeks) (Experimental): In Part A, HCV GT3-infected NC TN participants will take grazoprevir (100 mg) + uprifosbuvir (450 mg) + elbasvir (50 mg) q.d. by mouth for 8 weeks. Part A participants who relapsed following completion of therapy were offered the option of retreatment with 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d. and RBV (weight-based dosing) b.i.d. by mouth for 16 weeks during Part C.
  Interventions: Drug: Grazoprevir; Drug: Uprifosbuvir; Drug: Elbasvir; Drug: MK-3682B; Drug: Ribavirin (RBV)
- A4/B4: GT3 NC TN Grazoprevir+Uprifosbuvir+Ruzasvir (8 weeks) (Experimental): Participants will be randomized to either Part A or Part B. In Part A, HCV GT3-infected NC TN participants will take grazoprevir (100 mg) + uprifosbuvir (450 mg) + ruzasvir (60 mg) q.d. by mouth for 8 weeks. In Part B, HCV GT3-infected NC TN participants will take 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d. by mouth for 8 weeks. Part A participants who relapsed following completion of therapy were offered the option of retreatment with 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d. and RBV (weight-based dosing) b.i.d. by mouth for 16 weeks during Part C.
  Interventions: Drug: Grazoprevir; Drug: Uprifosbuvir; Drug: Ruzasvir; Drug: MK-3682B; Drug: Ribavirin (RBV)
- B5: GT3 NC TN MK-3682B + RBV (8 weeks) (Experimental): In Part B, HCV GT3-infected NC TN participants will take 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d., and RBV (weight-based dosing) b.i.d., by mouth for 8 weeks.
  Interventions: Drug: MK-3682B; Drug: Ribavirin (RBV)
- B6: GT3 NC TN MK-3682B (12 weeks) (Experimental): In Part B, HCV GT3-infected NC TN participants will take 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d. by mouth for 12 weeks.
  Interventions: Drug: MK-3682B
- B7: GT3 NC TN MK-3682B + RBV (12 weeks) (Experimental): In Part B, HCV GT3-infected NC TN participants will take 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d., and RBV (weight-based dosing) b.i.d., by mouth for 12 weeks.
  Interventions: Drug: MK-3682B; Drug: Ribavirin (RBV)
- B8: GT3 NC TE MK-3682B (8 weeks) (Experimental): In Part B, HCV GT3-infected NC TE participants will take 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d. by mouth for 8 weeks.
  Interventions: Drug: MK-3682B
- B9: GT3 NC TE MK-3682B + RBV (8 weeks) (Experimental): In Part B, HCV GT3-infected NC TE participants will take 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d., and RBV (weight-based dosing) b.i.d., by mouth for 8 weeks.
  Interventions: Drug: MK-3682B; Drug: Ribavirin (RBV)
- B10: GT3 NC TE MK-3682B (12 weeks) (Experimental): In Part B, HCV GT3-infected NC TE participants will take 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d. by mouth for 12 weeks.
  Interventions: Drug: MK-3682B
- B11: GT3 NC TE MK-3682B + RBV (12 weeks) (Experimental): In Part B, HCV GT3-infected NC TE participants will take 2 MK-3682 FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d., and RBV (weight-based dosing) b.i.d., by mouth for 12 weeks.
  Interventions: Drug: MK-3682B; Drug: Ribavirin (RBV)
- B12: GT3 NC TE MK-3682B (16 weeks) (Experimental): In Part B, HCV GT3-infected NC TE participants will take 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d. by mouth for 16 weeks.
  Interventions: Drug: MK-3682B
- B13: GT3 C TN MK-3682B (12 weeks) (Experimental): In Part B, HCV GT3-infected C TN participants will take 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d. by mouth for 12 weeks.
  Interventions: Drug: MK-3682B
- B14: GT3 C TN MK-3682B + RBV (12 weeks) (Experimental): In Part B, HCV GT3-infected C TN participants will take 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d., and RBV (weight-based dosing) b.i.d., by mouth for 12 weeks.
  Interventions: Drug: MK-3682B; Drug: Ribavirin (RBV)
- B15: GT3 C TN MK-3682B (16 weeks) (Experimental): In Part B, HCV GT3-infected C TN participants will take 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d. by mouth for 16 weeks.
  Interventions: Drug: MK-3682B
- B16: GT3 C TE MK-3682B (12 weeks) (Experimental): In Part B, HCV GT3-infected C TE participants will take 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d. by mouth for 12 weeks.
  Interventions: Drug: MK-3682B
- B17: GT3 C TE MK-3682B + RBV (12 weeks) (Experimental): In Part B, HCV GT3-infected C TE participants will take 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d., and RBV (weight-based dosing) b.i.d., by mouth for 12 weeks.
  Interventions: Drug: MK-3682B; Drug: Ribavirin (RBV)
- B18: GT3 C TE MK-3682B (16 weeks) (Experimental): In Part B, HCV GT3-infected C TE participants will take 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d. by mouth for 16 weeks.
  Interventions: Drug: MK-3682B
- B19: GT3 C TE MK-3682B + RBV (16 weeks) (Experimental): In Part B, HCV GT3-infected C TE participants will take 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d., and RBV (weight-based dosing) b.i.d., by mouth for 16 weeks.
  Interventions: Drug: MK-3682B; Drug: Ribavirin (RBV)
- B20: GT4 NC TN MK-3682B (8 weeks) (Experimental): In Part B, HCV GT4-infected NC TN participants will take 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d. by mouth for 8 weeks.
  Interventions: Drug: MK-3682B
- B21: GT5 NC TN MK-3682B (12 weeks) (Experimental): In Part B, HCV GT5-infected NC TN participants will take 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d. by mouth for 12 weeks.
  Interventions: Drug: MK-3682B
- B22: GT6 NC TN MK-3682B (12 weeks) (Experimental): In Part B, HCV GT6-infected NC TN participants will take 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d. by mouth for 12 weeks.
  Interventions: Drug: MK-3682B

INTERVENTIONS:
Drug: Grazoprevir — Part A: one grazoprevir 100 mg tablet taken q.d. by mouth.
  Other Names: MK-5172
  Arms: A1: GT3 NC TN Grazoprevir+Uprifosbuvir+Elbasvir (8 weeks); A2: GT3 NC TN Grazoprevir+Uprifosbuvir+Ruzasvir (8 weeks); A3: GT3 NC TN Grazoprevir+Uprifosbuvir+Elbasvir (8 weeks); A4/B4: GT3 NC TN Grazoprevir+Uprifosbuvir+Ruzasvir (8 weeks)
Drug: Uprifosbuvir — Part A: two or three uprifosbuvir 150 mg (300 or 450 mg total daily dose) tablets taken q.d. by mouth.
  Other Names: MK-3682
  Arms: A1: GT3 NC TN Grazoprevir+Uprifosbuvir+Elbasvir (8 weeks); A2: GT3 NC TN Grazoprevir+Uprifosbuvir+Ruzasvir (8 weeks); A3: GT3 NC TN Grazoprevir+Uprifosbuvir+Elbasvir (8 weeks); A4/B4: GT3 NC TN Grazoprevir+Uprifosbuvir+Ruzasvir (8 weeks)
Drug: Elbasvir — Part A: one elbasvir 50 mg tablet taken q.d. by mouth.
  Other Names: MK-8742
  Arms: A1: GT3 NC TN Grazoprevir+Uprifosbuvir+Elbasvir (8 weeks); A3: GT3 NC TN Grazoprevir+Uprifosbuvir+Elbasvir (8 weeks)
Drug: Ruzasvir — Part A: six ruzasvir 10 mg (60 mg total daily dose) capsules taken q.d. by mouth.
  Other Names: MK-8408
  Arms: A2: GT3 NC TN Grazoprevir+Uprifosbuvir+Ruzasvir (8 weeks); A4/B4: GT3 NC TN Grazoprevir+Uprifosbuvir+Ruzasvir (8 weeks)
Drug: MK-3682B — Part B and Part C: two FDC tablets, each containing grazoprevir 50 mg + elbasvir 225 mg + ruzasvir 30 mg, taken q.d. by mouth.
Drug: Ribavirin (RBV) — Part B and Part C: RBV 200 mg capsules taken b.i.d. by mouth at a total daily dose of 800 mg - 1400 mg based on participant body weight.
  Other Names: Rebetol
  Arms: A1: GT3 NC TN Grazoprevir+Uprifosbuvir+Elbasvir (8 weeks); A2: GT3 NC TN Grazoprevir+Uprifosbuvir+Ruzasvir (8 weeks); A3: GT3 NC TN Grazoprevir+Uprifosbuvir+Elbasvir (8 weeks); A4/B4: GT3 NC TN Grazoprevir+Uprifosbuvir+Ruzasvir (8 weeks); B11: GT3 NC TE MK-3682B + RBV (12 weeks); B14: GT3 C TN MK-3682B + RBV (12 weeks); B17: GT3 C TE MK-3682B + RBV (12 weeks); B19: GT3 C TE MK-3682B + RBV (16 weeks); B5: GT3 NC TN MK-3682B + RBV (8 weeks); B7: GT3 NC TN MK-3682B + RBV (12 weeks); B9: GT3 NC TE MK-3682B + RBV (8 weeks)

SUMMARY:
This is a randomized, three-part, parallel-group, open-label trial of grazoprevir (MK-5172) (100 mg) and uprifosbuvir (MK-3682) (300 mg or 450 mg) with either elbasvir (MK-8742) (50 mg) or ruzasvir (MK-8408) (60 mg), and with or without ribavirin (RBV), in treatment-naive (TN) or treatment-experienced (TE) cirrhotic (C) or non-cirrhotic (NC) participants infected with hepatitis C virus (HCV) genotype (GT) 3, GT4, GT5, or GT6. Part A will consist of 4 arms to evaluate the safety of dose combinations. In Part B, participants will take 2 uprifosbuvir (+) grazoprevir (+) ruzasvir (MK-3682B) fixed dose combination (FDC) tablets once daily (q.d.) by mouth, with or without twice-daily (b.i.d.) RBV (200 mg capsules; weight-based dosing). Participants who relapse following completion of therapy in Part A will be offered the option of retreatment with 16 weeks of uprifosbuvir (+) grazoprevir (+) ruzasvir with RBV in Part C (data obtained from Part C will not be used in the analysis of outcome measures).

DETAILED DESCRIPTION:
In Part A, study therapy will be administered as separate products, each taken q.d. by mouth. In Part B and Part C, participants will take 2 uprifosbuvir (+) grazoprevir (+) ruzasvir FDC tablets q.d. by mouth; each uprifosbuvir (+) grazoprevir (+) ruzasvir FDC tablet contains grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg.

ELIGIBILITY:
Inclusion Criteria:

* Has documented chronic HCV GT3, GT4, GT5, or GT6 with no evidence of non-typeable or mixed GT infection
* Is otherwise healthy as determined by the medical history, physical examination, electrocardiogram (ECG), and clinical laboratory measurements performed at the time of screening
* Has cirrhosis of the liver (Part B only) or is non-cirrhotic (Part A and B)
* Is HCV treatment-naïve or has experienced virologic failure after completing a prior Pegylated Interferon/Ribavirin (Peg-IFN/RBV) regimen
* Is of non childbearing potential or agrees to avoid becoming pregnant or impregnating a partner beginning at least 2 weeks prior to administration of the initial dose of study drug and for 14 days after the last dose of study drug if not taking RBV, or for 6 months after the last dose of study drug if taking RBV (or longer if dictated by local regulations). If not abstinent from heterosexual activity, participants in Part A must use 2 acceptable forms of barrier contraception whereas participants in Parts B and C must use 2 acceptable forms of contraception which may include oral contraceptives

Part B only:

* If coinfected with human immunodeficiency virus (HIV) is not currently on antiretroviral therapy (ART) and has no plans to initiate ART treatment while participating in this study OR has well-controlled HIV on ART.
* Has at least 1 viable antiretroviral regimen alternative beyond their current regimen in the event of HIV virologic failure and the development of anti-retroviral drug resistance.

Exclusion Criteria:

Parts A, B, and C (unless otherwise specified):

* Has evidence of decompensated liver disease manifested by the presence of or history of ascites, esophageal or gastric variceal bleeding, hepatic encephalopathy or other signs or symptoms of advanced liver disease.
* If cirrhotic (Part B only), is Child-Pugh Class B or C or has a Pugh-Turcotte (CPT) score >5.
* Is coinfected with hepatitis B virus (Parts A, B, and C) or is coinfected with HIV (Part A only; HIV coinfected participants are eligible for Parts B and C).
* If coinfected with HIV, has a history of opportunistic infection in the preceding 6 months prior to screening.
* Has a history of malignancy ≤5 years prior to signing informed consent except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer or carcinoma in situ; or is under evaluation for other active or suspected malignancy.
* Has cirrhosis and liver imaging within 6 months of Day 1 showing evidence of hepatocellular carcinoma (HCC) or is under evaluation for HCC.
* Has clinically-relevant drug or alcohol abuse within 12 months of screening.
* Is female and is pregnant or breastfeeding, or expecting to conceive or donate eggs from at least 2 weeks prior to Day 1 and 6 months after the last dose of study medication, or longer if dictated by local regulations OR a male participant who is expecting to donate sperm from at least 2 weeks prior to day 1 until 6 months after the last dose of study medication.
* Has any of the following conditions:
* Organ transplants (including hematopoietic stem cell transplants) other than cornea and hair.
* Poor venous access that precludes routine peripheral blood sampling required for this trial.
* History of gastric surgery (e.g., stapling, bypass) or a history of malabsorption disorders (e.g., celiac sprue disease).
* Current or history of any clinically significant cardiac abnormalities/dysfunction, including but not limited to: angina, congestive heart failure, myocardial infarction, pulmonary hypertension, complex congenital heart disease, cardiomyopathy, significant arrhythmia, uncontrolled hypertension, a history of use of antianginal or anti-arrythmic agents for cardiac conditions, prolonged ECG QTc interval (>470 ms for males or >480 ms for females by either the Fridericia formula) at the screening visit, personal or family history of Torsade de pointes.
* Chronic pulmonary disease, including but not limited to: clinically significant chronic obstructive pulmonary disease, interstitial lung disease, pulmonary fibrosis, sarcoidosis.
* Central nervous system (CNS) trauma requiring intubation, intracranial pressure monitoring, brain meningeal or skull surgery, or resulting in seizure, coma, permanent neurologic deficits, abnormal brain imaging, or cerebral spinal fluid (CSF) leak. Prior brain hemorrhage and/or intracranial aneurysms (whether adequately repaired or not).
* Current or history of seizure disorder unless seizure was >10 years ago, a single isolated event, no history of or current use of anti-seizure medications prescribed, and a normal neurological examination is documented in trial files within 6 months of Day 1.
* Has a history of stroke or transient ischemic attack.
* Has a history of a medical/surgical condition that resulted in hospitalization within the 3 months prior to enrollment, other than for minor elective procedures.
* Has medical/surgical conditions that may result in a need for hospitalization during the period of the study.
* Has any medical condition requiring, or likely to require, chronic systemic administration of corticosteroids, tumor necrosis factor (TNF) antagonists, or other immunosuppressant drugs during the course of the trial.
* Has any condition, prestudy laboratory or ECG abnormality or history of any illness, which, in the opinion of the investigator, might confound the results of the study or pose additional risk in administering the study drugs to the participant.
* Has had a life-threatening serious adverse event (SAE) during the screening period.
* Has evidence of history of chronic hepatitis not caused by HCV, including but not limited to nonalcoholic steatohepatitis (NASH), drug-induced hepatitis, hemochromatosis, Wilson's disease, α1-antitrypsin deficiency, alcoholic liver disease and autoimmune hepatitis Parts B and C only: is a male whose female partner(s) is/are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 413 (Actual)
Dates: Start 2015-01-28 (Actual); Primary Completion 2016-09-19 (Actual); Study Completion 2017-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Lawitz E, Buti M, Vierling JM, Almasio PL, Bruno S, Ruane PJ, Hassanein TI, Muellhaupt B, Pearlman B, Jancoriene L, Gao W, Huang HC, Shepherd A, Tannenbaum B, Fernsler D, Li JJ, Grandhi A, Liu H, Su FH, Wan S, Dutko FJ, Nguyen BT, Wahl J, Robertson MN, Barr E, Yeh WW, Plank RM, Butterton JR, Yoshida EM. Safety and efficacy of a fixed-dose combination regimen of grazoprevir, ruzasvir, and uprifosbuvir with or without ribavirin in participants with and without cirrhosis with chronic hepatitis C virus genotype 1, 2, or 3 infection (C-CREST-1 and C-CREST-2, part B): two randomised, phase 2, open-label trials. Lancet Gastroenterol Hepatol. 2017 Nov;2(11):814-823. doi: 10.1016/S2468-1253(17)30163-2. Epub 2017 Aug 10. PMID 28802814
- [Derived] Gane EJ, Pianko S, Roberts SK, Thompson AJ, Zeuzem S, Zuckerman E, Ben-Ari Z, Foster GR, Agarwal K, Laursen AL, Gerstoft J, Gao W, Huang HC, Fitzgerald B, Fernsler D, Li JJ, Grandhi A, Liu H, Su FH, Wan S, Zeng Z, Chen HL, Dutko FJ, Nguyen BT, Wahl J, Robertson MN, Barr E, Yeh WW, Plank RM, Butterton JR, Esteban R. Safety and efficacy of an 8-week regimen of grazoprevir plus ruzasvir plus uprifosbuvir compared with grazoprevir plus elbasvir plus uprifosbuvir in participants without cirrhosis infected with hepatitis C virus genotypes 1, 2, or 3 (C-CREST-1 and C-CREST-2, part A): two randomised, phase 2, open-label trials. Lancet Gastroenterol Hepatol. 2017 Nov;2(11):805-813. doi: 10.1016/S2468-1253(17)30159-0. Epub 2017 Aug 10. PMID 28802816

RESULTS

PARTICIPANT FLOW:
Recruitment Details: No participants were randomized to the 'B21: GT5 NC TN MK-3682B (12 weeks)' arm.
Pre-assignment Details: Participants were enrolled into either Part A or Part B. Part A enrolled non-cirrhotic (NC), treatment-naïve (TN) participants with hepatitis C virus (HCV) genotype (GT) 3; Part B enrolled NC or cirrhotic (C), TN or treatment-experienced (TE) participants with HCV GT3, GT4, GT5 or GT6. Participants who relapsed in Part A were retreated in Part C.
Groups:
- A1: GT3 NC TN Grazoprevir+Uprifosbuvir+Elbasvir (8 Weeks): In Part A, HCV GT3-infected NC TN participants received grazoprevir (100 mg) + uprifosbuvir (300 mg) + elbasvir (50 mg) q.d. by mouth for 8 weeks. Part A participants who relapsed following completion of therapy were offered the option of retreatment with 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d. and RBV (weight-based dosing) b.i.d. by mouth for 16 weeks during Part C.
- A2: GT3 NC TN Grazoprevir+Uprifosbuvir+Ruzasvir (8 Weeks): In Part A, HCV GT3-infected NC TN participants received grazoprevir (100 mg) + uprifosbuvir (300 mg) + ruzasvir (60 mg) q.d. by mouth for 8 weeks. Part A participants who relapsed following completion of therapy were offered the option of retreatment with 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d. and RBV (weight-based dosing) b.i.d. by mouth for 16 weeks during Part C.
- A3: GT3 NC TN Grazoprevir+Uprifosbuvir+Elbasvir (8 Weeks): In Part A, HCV GT3-infected NC TN participants received grazoprevir (100 mg) + uprifosbuvir (450 mg) + elbasvir (50 mg) q.d. by mouth for 8 weeks. Part A participants who relapsed following completion of therapy were offered the option of retreatment with 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d. and RBV (weight-based dosing) b.i.d. by mouth for 16 weeks during Part C.
- A4: GT3 NC TN Grazoprevir+Uprifosbuvir+Ruzasvir (8 Weeks): In Part A, HCV GT3-infected NC TN participants received grazoprevir 100 mg + uprifosbuvir 450 mg + ruzasvir 60 mg q.d. by mouth for 8 weeks. Part A participants who relapsed following completion of therapy received retreatment with 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d. and RBV (weight-based dosing) b.i.d. by mouth for 16 weeks during Part C.
- B4: GT3 NC TN MK-3682B (8 Weeks): In Part B, HCV GT3-infected NC TN participants received 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d. by mouth for 8 weeks.
- B5: GT3 NC TN MK-3682B + RBV (8 Weeks): In Part B, HCV GT3-infected NC TN participants received 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d., and RBV (weight-based dosing) b.i.d., by mouth for 8 weeks.
- B6: GT3 NC TN MK-3682B (12 Weeks): In Part B, HCV GT3-infected NC TN participants received 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d. by mouth for 12 weeks.
- B7: GT3 NC TN MK-3682B + RBV (12 Weeks): In Part B, HCV GT3-infected NC TN participants received 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d., and RBV (weight-based dosing) b.i.d., by mouth for 12 weeks.
- B8: GT3 NC TE MK-3682B (8 Weeks): In Part B, HCV GT3-infected NC TE participants received 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d. by mouth for 8 weeks.
- B9: GT3 NC TE MK-3682B + RBV (8 Weeks): In Part B, HCV GT3-infected NC TE participants received 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d., and RBV (weight-based dosing) b.i.d., by mouth for 8 weeks.
- B10: GT3 NC TE MK-3682B (12 Weeks): In Part B, HCV GT3-infected NC TE participants received 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d. by mouth for 12 weeks.
- B11: GT3 NC TE MK-3682B + RBV (12 Weeks): In Part B, HCV GT3-infected NC TE participants received 2 MK-3682 FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d., and RBV (weight-based dosing) b.i.d., by mouth for 12 weeks.
- B12: GT3 NC TE MK-3682B (16 Weeks): In Part B, HCV GT3-infected NC TE participants received 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d. by mouth for 16 weeks.
- B13: GT3 C TN MK-3682B (12 Weeks): In Part B, HCV GT3-infected C TN participants received 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d. by mouth for 12 weeks.
- B14: GT3 C TN MK-3682B + RBV (12 Weeks): In Part B, HCV GT3-infected C TN participants received 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d., and RBV (weight-based dosing) b.i.d., by mouth for 12 weeks.
- B15: GT3 C TN MK-3682B (16 Weeks): In Part B, HCV GT3-infected C TN participants received 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d. by mouth for 16 weeks.
- B16: GT3 C TE MK-3682B (12 Weeks): In Part B, HCV GT3-infected C TE participants received 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d. by mouth for 12 weeks.
- B17: GT3 C TE MK-3682B + RBV (12 Weeks): In Part B, HCV GT3-infected C TE participants received 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d., and RBV (weight-based dosing) b.i.d., by mouth for 12 weeks.
- B18: GT3 C TE MK-3682B (16 Weeks): In Part B, HCV GT3-infected C TE participants received 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d. by mouth for 16 weeks.
- B19: GT3 C TE MK-3682B + RBV (16 Weeks): In Part B, HCV GT3-infected C TE participants received 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d., and RBV (weight-based dosing) b.i.d., by mouth for 16 weeks.
- B20: GT4 NC TN MK-3682B (8 Weeks): In Part B, HCV GT4-infected NC TN participants received 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d. by mouth for 8 weeks.
- B21: GT5 NC TN MK-3682B (12 Weeks): In Part B, HCV GT5-infected NC TN participants received 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d. by mouth for 12 weeks.
- B22: GT6 NC TN MK-3682B (12 Weeks): In Part B, HCV GT6-infected NC TN participants received 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d. by mouth for 12 weeks.
Period: Part A and Part B
Arm/Group | A1: GT3 NC TN Grazoprevir+Uprifosbuvir+Elbasvir (8 Weeks) | A2: GT3 NC TN Grazoprevir+Uprifosbuvir+Ruzasvir (8 Weeks) | A3: GT3 NC TN Grazoprevir+Uprifosbuvir+Elbasvir (8 Weeks) | A4: GT3 NC TN Grazoprevir+Uprifosbuvir+Ruzasvir (8 Weeks) | B4: GT3 NC TN MK-3682B (8 Weeks) | B5: GT3 NC TN MK-3682B + RBV (8 Weeks) | B6: GT3 NC TN MK-3682B (12 Weeks) | B7: GT3 NC TN MK-3682B + RBV (12 Weeks) | B8: GT3 NC TE MK-3682B (8 Weeks) | B9: GT3 NC TE MK-3682B + RBV (8 Weeks) | B10: GT3 NC TE MK-3682B (12 Weeks) | B11: GT3 NC TE MK-3682B + RBV (12 Weeks) | B12: GT3 NC TE MK-3682B (16 Weeks) | B13: GT3 C TN MK-3682B (12 Weeks) | B14: GT3 C TN MK-3682B + RBV (12 Weeks) | B15: GT3 C TN MK-3682B (16 Weeks) | B16: GT3 C TE MK-3682B (12 Weeks) | B17: GT3 C TE MK-3682B + RBV (12 Weeks) | B18: GT3 C TE MK-3682B (16 Weeks) | B19: GT3 C TE MK-3682B + RBV (16 Weeks) | B20: GT4 NC TN MK-3682B (8 Weeks) | B21: GT5 NC TN MK-3682B (12 Weeks) | B22: GT6 NC TN MK-3682B (12 Weeks)
Started | 21 | 21 | 22 | 22 | 16 | 36 | 37 | 35 | 15 | 14 | 14 | 15 | 16 | 13 | 16 | 14 | 15 | 14 | 21 | 25 | 7 | 0 | 4
Treated | 21 | 21 | 22 | 22 | 16 | 36 | 37 | 35 | 15 | 14 | 14 | 15 | 16 | 13 | 16 | 14 | 15 | 14 | 20 | 25 | 7 | 0 | 4
Completed | 20 | 21 | 22 | 22 | 16 | 33 | 36 | 34 | 15 | 14 | 14 | 15 | 16 | 13 | 16 | 13 | 15 | 13 | 20 | 24 | 7 | 0 | 4
Not Completed | 1 | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Period: Part C
Arm/Group | A1: GT3 NC TN Grazoprevir+Uprifosbuvir+Elbasvir (8 Weeks) | A2: GT3 NC TN Grazoprevir+Uprifosbuvir+Ruzasvir (8 Weeks) | A3: GT3 NC TN Grazoprevir+Uprifosbuvir+Elbasvir (8 Weeks) | A4: GT3 NC TN Grazoprevir+Uprifosbuvir+Ruzasvir (8 Weeks) | B4: GT3 NC TN MK-3682B (8 Weeks) | B5: GT3 NC TN MK-3682B + RBV (8 Weeks) | B6: GT3 NC TN MK-3682B (12 Weeks) | B7: GT3 NC TN MK-3682B + RBV (12 Weeks) | B8: GT3 NC TE MK-3682B (8 Weeks) | B9: GT3 NC TE MK-3682B + RBV (8 Weeks) | B10: GT3 NC TE MK-3682B (12 Weeks) | B11: GT3 NC TE MK-3682B + RBV (12 Weeks) | B12: GT3 NC TE MK-3682B (16 Weeks) | B13: GT3 C TN MK-3682B (12 Weeks) | B14: GT3 C TN MK-3682B + RBV (12 Weeks) | B15: GT3 C TN MK-3682B (16 Weeks) | B16: GT3 C TE MK-3682B (12 Weeks) | B17: GT3 C TE MK-3682B + RBV (12 Weeks) | B18: GT3 C TE MK-3682B (16 Weeks) | B19: GT3 C TE MK-3682B + RBV (16 Weeks) | B20: GT4 NC TN MK-3682B (8 Weeks) | B21: GT5 NC TN MK-3682B (12 Weeks) | B22: GT6 NC TN MK-3682B (12 Weeks)
Started | 2 (Part A participants who had relapsed were offered the option of retreatment in Part C.) | 1 (Part A participants who had relapsed were offered the option of retreatment in Part C.) | 3 (Part A participants who had relapsed were offered the option of retreatment in Part C.) | 2 (Part A participants who had relapsed were offered the option of retreatment in Part C.) | 0 (Part B participants were not included in Part C.) | 0 (Part B participants were not included in Part C.) | 0 (Part B participants were not included in Part C.) | 0 (Part B participants were not included in Part C.) | 0 (Part B participants were not included in Part C.) | 0 (Part B participants were not included in Part C.) | 0 (Part B participants were not included in Part C.) | 0 (Part B participants were not included in Part C.) | 0 (Part B participants were not included in Part C.) | 0 (Part B participants were not included in Part C.) | 0 (Part B participants were not included in Part C.) | 0 (Part B participants were not included in Part C.) | 0 (Part B participants were not included in Part C.) | 0 (Part B participants were not included in Part C.) | 0 (Part B participants were not included in Part C.) | 0 (Part B participants were not included in Part C.) | 0 (Part B participants were not included in Part C.) | 0 | 0 (Part B participants were not included in Part C.)
Completed | 2 | 1 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Overall Number of Baseline Participants includes participants who received at least one dose of study drug. One 'B18: GT3 C TE MK-3682B (16 weeks)' participant did not receive any study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | A1: GT3 NC TN Grazoprevir+Uprifosbuvir+Elbasvir (8 Weeks) | A2: GT3 NC TN Grazoprevir+Uprifosbuvir+Ruzasvir (8 Weeks) | A3: GT3 NC TN Grazoprevir+Uprifosbuvir+Elbasvir (8 Weeks) | A4: GT3 NC TN Grazoprevir+Uprifosbuvir+Ruzasvir (8 Weeks) | B4: GT3 NC TN MK-3682B (8 Weeks) | B5: GT3 NC TN MK-3682B + RBV (8 Weeks) | B6: GT3 NC TN MK-3682B (12 Weeks) | B7: GT3 NC TN MK-3682B + RBV (12 Weeks) | B8: GT3 NC TE MK-3682B (8 Weeks) | B9: GT3 NC TE MK-3682B + RBV (8 Weeks) | B10: GT3 NC TE MK-3682B (12 Weeks) | B11: GT3 NC TE MK-3682B + RBV (12 Weeks) | B12: GT3 NC TE MK-3682B (16 Weeks) | B13: GT3 C TN MK-3682B (12 Weeks) | B14: GT3 C TN MK-3682B + RBV (12 Weeks) | B15: GT3 C TN MK-3682B (16 Weeks) | B16: GT3 C TE MK-3682B (12 Weeks) | B17: GT3 C TE MK-3682B + RBV (12 Weeks) | B18: GT3 C TE MK-3682B (16 Weeks) | B19: GT3 C TE MK-3682B + RBV (16 Weeks) | B20: GT4 NC TN MK-3682B (8 Weeks) | B21: GT5 NC TN MK-3682B (12 Weeks) | B22: GT6 NC TN MK-3682B (12 Weeks) | Total
Number analyzed (Participants) | 21 | 21 | 22 | 22 | 16 | 36 | 37 | 35 | 15 | 14 | 14 | 15 | 16 | 13 | 16 | 14 | 15 | 14 | 20 | 25 | 7 | 0 | 4 | 412
Age, Customized [Number; unit: Participants]
  Less than 18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0
  18 to 35 years | 4 | 4 | 3 | 4 | 3 | 8 | 9 | 7 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 |  | 0 | 49
  36 to 50 years | 12 | 9 | 14 | 12 | 4 | 11 | 14 | 12 | 5 | 5 | 6 | 4 | 6 | 7 | 3 | 3 | 4 | 3 | 6 | 6 | 3 |  | 1 | 150
  51 to 64 years | 5 | 8 | 5 | 3 | 6 | 16 | 13 | 16 | 8 | 7 | 6 | 9 | 9 | 4 | 13 | 9 | 11 | 9 | 13 | 18 | 3 |  | 3 | 194
  Over 64 years | 0 | 0 | 0 | 3 | 3 | 1 | 1 | 0 | 2 | 1 | 0 | 1 | 1 | 2 | 0 | 2 | 0 | 0 | 1 | 1 | 0 |  | 0 | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 15 | 14 | 11 | 7 | 19 | 23 | 23 | 7 | 2 | 8 | 6 | 5 | 3 | 5 | 3 | 8 | 1 | 2 | 5 | 1 |  | 2 | 179
  Male | 12 | 6 | 8 | 11 | 9 | 17 | 14 | 12 | 8 | 12 | 6 | 9 | 11 | 10 | 11 | 11 | 7 | 13 | 18 | 20 | 6 |  | 2 | 233

OUTCOME MEASURES:

1. Primary Outcome: Percentage of HCV GT3-infected Participants Achieving Sustained Virologic Response at Follow-up Week 12 (SVR12)
Description: SVR12 is defined as HCV ribonucleic acid (RNA) less than the lower limit of quantification (<LLOQ, 15 IU/mL) 12 weeks after the end of all study therapy. A4+B4: GT3 NC TN MK-3682B (8 weeks) arm includes both participants from Part A and Part B who received equivalent dose of MK-3682B.
Time Frame: Up to 20 weeks (Part A), up to 28 weeks (Part B)
Population: Analysis population included HCV GT3 participants who received treatment and did not have major protocol deviations that may substantially affect the results of the SVR endpoints. Therefore, only GT3 treatment arms are presented in the table below.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- A1: GT3 NC TN Grazoprevir+Uprifosbuvir+Elbasvir (8 Weeks): In Part A, HCV GT3-infected NC TN participants received grazoprevir (100 mg) + uprifosbuvir (300 mg) + elbasvir (50 mg) q.d. by mouth for 8 weeks.
- A2: GT3 NC TN Grazoprevir+Uprifosbuvir+Ruzasvir (8 Weeks): In Part A, HCV GT3-infected NC TN participants received grazoprevir (100 mg) + uprifosbuvir (300 mg) + ruzasvir (60 mg) q.d. by mouth for 8 weeks.
- A3: GT3 NC TN Grazoprevir+Uprifosbuvir+Elbasvir (8 Weeks): In Part A, HCV GT3-infected NC TN participants received grazoprevir (100 mg) + uprifosbuvir (450 mg) + elbasvir (50 mg) q.d. by mouth for 8 weeks.
- A4: GT3 NC TN Grazoprevir+Uprifosbuvir+Ruzasvir (8 Weeks): In Part A, HCV GT3-infected NC TN participants received grazoprevir 100 mg + uprifosbuvir 450 mg + ruzasvir 60 mg q.d. by mouth for 8 weeks.
- A4+B4: GT3 NC TN MK-3682B (8 Weeks): HCV GT3-infected NC TN participants received grazoprevir 100 mg + uprifosbuvir 450 mg + ruzasvir 60 mg q.d. by mouth for 8 weeks during Part A or 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d. by mouth for 8 weeks during Part B.
- B4: GT3 NC TN MK-3682B (8 Weeks): HCV GT3-infected NC TN participants received 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d. by mouth for 8 weeks during Part B
Arm/Group | A1: GT3 NC TN Grazoprevir+Uprifosbuvir+Elbasvir (8 Weeks) | A2: GT3 NC TN Grazoprevir+Uprifosbuvir+Ruzasvir (8 Weeks) | A3: GT3 NC TN Grazoprevir+Uprifosbuvir+Elbasvir (8 Weeks) | A4: GT3 NC TN Grazoprevir+Uprifosbuvir+Ruzasvir (8 Weeks) | A4+B4: GT3 NC TN MK-3682B (8 Weeks) | B4: GT3 NC TN MK-3682B (8 Weeks) | B5: GT3 NC TN MK-3682B + RBV (8 Weeks) | B6: GT3 NC TN MK-3682B (12 Weeks) | B7: GT3 NC TN MK-3682B + RBV (12 Weeks) | B8: GT3 NC TE MK-3682B (8 Weeks) | B9: GT3 NC TE MK-3682B + RBV (8 Weeks) | B10: GT3 NC TE MK-3682B (12 Weeks) | B11: GT3 NC TE MK-3682B + RBV (12 Weeks) | B12: GT3 NC TE MK-3682B (16 Weeks) | B13: GT3 C TN MK-3682B (12 Weeks) | B14: GT3 C TN MK-3682B + RBV (12 Weeks) | B15: GT3 C TN MK-3682B (16 Weeks) | B16: GT3 C TE MK-3682B (12 Weeks) | B17: GT3 C TE MK-3682B + RBV (12 Weeks) | B18: GT3 C TE MK-3682B (16 Weeks) | B19: GT3 C TE MK-3682B + RBV (16 Weeks)
Number analyzed (Participants) | 21 | 21 | 22 | 22 | 38 | 16 | 35 | 36 | 35 | 15 | 14 | 14 | 15 | 16 | 13 | 16 | 13 | 15 | 14 | 20 | 25
Percentage of participants | 90.5 [69.6 to 98.8] | 95.2 [76.2 to 99.9] | 86.4 [65.1 to 97.1] | 90.9 [70.8 to 98.9] | 92.1 [78.6 to 98.3] | 93.8 [69.8 to 99.8] | 100.0 [90.0 to 100.0] | 97.2 [85.5 to 99.9] | 100.0 [90.0 to 100.0] | 100.0 [78.2 to 100.0] | 92.9 [66.1 to 99.8] | 100.0 [76.8 to 100.0] | 93.3 [68.1 to 99.8] | 93.8 [69.8 to 99.8] | 92.3 [64.0 to 99.8] | 100.0 [79.4 to 100.0] | 100.0 [75.3 to 100.0] | 100.0 [78.2 to 100.0] | 100.0 [76.8 to 100.0] | 100.0 [83.2 to 100.0] | 96.0 [79.6 to 99.9]

2. Primary Outcome: Number of Participants Experiencing an Adverse Event (AE)
Description: An adverse event is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. Part C in the table below combines all (eight) participants from the four distinct arms of Part A who relapsed and were subsequently treated with MK-3682B + RBV for 16 weeks.
Time Frame: Up to 40 weeks
Population: All participants who received at least 1 dose of study drug, categorized according to the treatment actually received. A4+B4 arm includes both participants from Part A and Part B who received equivalent dose of MK-3682B. Part C arm includes participants who relapsed following the completion of Part A therapy and received treatment during Part C.
Measure: Count of Participants; unit: Participants
Groups:
- A4+ B4: GT3 NC TN MK-3682B (8 Weeks): HCV GT3-infected NC TN participants received grazoprevir 100 mg + uprifosbuvir 450 mg + ruzasvir 60 mg q.d. by mouth for 8 weeks during Part A or 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d. by mouth for 8 weeks during Part B.
- Part C: GT3 NC TN: MK-3682B + RBV (16 Weeks): Part A participants who relapsed following completion of therapy were offered the option of retreatment with 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d. and RBV (weight-based dosing) b.i.d. by mouth for 16 weeks during Part C.
Arm/Group | A1: GT3 NC TN Grazoprevir+Uprifosbuvir+Elbasvir (8 Weeks) | A2: GT3 NC TN Grazoprevir+Uprifosbuvir+Ruzasvir (8 Weeks) | A3: GT3 NC TN Grazoprevir+Uprifosbuvir+Elbasvir (8 Weeks) | A4: GT3 NC TN Grazoprevir+Uprifosbuvir+Ruzasvir (8 Weeks) | A4+ B4: GT3 NC TN MK-3682B (8 Weeks) | B4: GT3 NC TN MK-3682B (8 Weeks) | B5: GT3 NC TN MK-3682B + RBV (8 Weeks) | B6: GT3 NC TN MK-3682B (12 Weeks) | B7: GT3 NC TN MK-3682B + RBV (12 Weeks) | B8: GT3 NC TE MK-3682B (8 Weeks) | B9: GT3 NC TE MK-3682B + RBV (8 Weeks) | B10: GT3 NC TE MK-3682B (12 Weeks) | B11: GT3 NC TE MK-3682B + RBV (12 Weeks) | B12: GT3 NC TE MK-3682B (16 Weeks) | B13: GT3 C TN MK-3682B (12 Weeks) | B14: GT3 C TN MK-3682B + RBV (12 Weeks) | B15: GT3 C TN MK-3682B (16 Weeks) | B16: GT3 C TE MK-3682B (12 Weeks) | B17: GT3 C TE MK-3682B + RBV (12 Weeks) | B18: GT3 C TE MK-3682B (16 Weeks) | B19: GT3 C TE MK-3682B + RBV (16 Weeks) | B20: GT4 NC TN MK-3682B (8 Weeks) | B22: GT6 NC TN MK-3682B (12 Weeks) | Part C: GT3 NC TN: MK-3682B + RBV (16 Weeks)
Number analyzed (Participants) | 21 | 21 | 22 | 22 | 38 | 16 | 36 | 37 | 35 | 15 | 14 | 14 | 15 | 16 | 13 | 16 | 14 | 15 | 14 | 20 | 25 | 7 | 4 | 8
Participants | 18 | 14 | 16 | 17 | 26 | 9 | 30 | 25 | 33 | 12 | 12 | 9 | 13 | 13 | 9 | 14 | 12 | 12 | 12 | 16 | 21 | 3 | 3 | 7

3. Primary Outcome: Number of Participants Who Had Study Drug Discontinued Due to an AE
Description: as for outcome 2
Time Frame: Up to 16 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | A1: GT3 NC TN Grazoprevir+Uprifosbuvir+Elbasvir (8 Weeks) | A2: GT3 NC TN Grazoprevir+Uprifosbuvir+Ruzasvir (8 Weeks) | A3: GT3 NC TN Grazoprevir+Uprifosbuvir+Elbasvir (8 Weeks) | A4: GT3 NC TN Grazoprevir+Uprifosbuvir+Ruzasvir (8 Weeks) | A4+ B4: GT3 NC TN MK-3682B (8 Weeks) | B4: GT3 NC TN MK-3682B (8 Weeks) | B5: GT3 NC TN MK-3682B + RBV (8 Weeks) | B6: GT3 NC TN MK-3682B (12 Weeks) | B7: GT3 NC TN MK-3682B + RBV (12 Weeks) | B8: GT3 NC TE MK-3682B (8 Weeks) | B9: GT3 NC TE MK-3682B + RBV (8 Weeks) | B10: GT3 NC TE MK-3682B (12 Weeks) | B11: GT3 NC TE MK-3682B + RBV (12 Weeks) | B12: GT3 NC TE MK-3682B (16 Weeks) | B13: GT3 C TN MK-3682B (12 Weeks) | B14: GT3 C TN MK-3682B + RBV (12 Weeks) | B15: GT3 C TN MK-3682B (16 Weeks) | B16: GT3 C TE MK-3682B (12 Weeks) | B17: GT3 C TE MK-3682B + RBV (12 Weeks) | B18: GT3 C TE MK-3682B (16 Weeks) | B19: GT3 C TE MK-3682B + RBV (16 Weeks) | B20: GT4 NC TN MK-3682B (8 Weeks) | B22: GT6 NC TN MK-3682B (12 Weeks) | Part C: GT3 NC TN: MK-3682B + RBV (16 Weeks)
Number analyzed (Participants) | 21 | 21 | 22 | 22 | 38 | 16 | 36 | 37 | 35 | 15 | 14 | 14 | 15 | 16 | 13 | 16 | 14 | 15 | 14 | 20 | 25 | 7 | 4 | 8
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0

4. Secondary Outcome: Percentage of GT3-infected Participants Achieving SVR at Follow-up Week 24 (SVR24)
Description: SVR24 is defined as HCV RNA <LLOQ of 15 IU/mL 24 weeks after the end of all study therapy. A4+B4: GT3 NC TN MK-3682B (8 weeks) arm includes both participants from Part A and Part B who received equivalent dose of MK-3682B.
Time Frame: Up to 40 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- A4+B4: GT3 NC TN MK-3682B (8 Weeks); B4: GT3 NC TN MK-3682B (8 Weeks): In Part B, HCV GT3-infected NC TN participants received 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d. by mouth for 8 weeks.
Arm/Group | A1: GT3 NC TN Grazoprevir+Uprifosbuvir+Elbasvir (8 Weeks) | A2: GT3 NC TN Grazoprevir+Uprifosbuvir+Ruzasvir (8 Weeks) | A3: GT3 NC TN Grazoprevir+Uprifosbuvir+Elbasvir (8 Weeks) | A4: GT3 NC TN Grazoprevir+Uprifosbuvir+Ruzasvir (8 Weeks) | A4+B4: GT3 NC TN MK-3682B (8 Weeks) | B4: GT3 NC TN MK-3682B (8 Weeks) | B5: GT3 NC TN MK-3682B + RBV (8 Weeks) | B6: GT3 NC TN MK-3682B (12 Weeks) | B7: GT3 NC TN MK-3682B + RBV (12 Weeks) | B8: GT3 NC TE MK-3682B (8 Weeks) | B9: GT3 NC TE MK-3682B + RBV (8 Weeks) | B10: GT3 NC TE MK-3682B (12 Weeks) | B11: GT3 NC TE MK-3682B + RBV (12 Weeks) | B12: GT3 NC TE MK-3682B (16 Weeks) | B13: GT3 C TN MK-3682B (12 Weeks) | B14: GT3 C TN MK-3682B + RBV (12 Weeks) | B15: GT3 C TN MK-3682B (16 Weeks) | B16: GT3 C TE MK-3682B (12 Weeks) | B17: GT3 C TE MK-3682B + RBV (12 Weeks) | B18: GT3 C TE MK-3682B (16 Weeks) | B19: GT3 C TE MK-3682B + RBV (16 Weeks)
Number analyzed (Participants) | 20 | 21 | 22 | 22 | 38 | 16 | 33 | 36 | 34 | 15 | 14 | 14 | 15 | 16 | 13 | 16 | 13 | 15 | 13 | 20 | 25
Percentage of participants | 90.0 [68.3 to 98.8] | 95.2 [76.2 to 99.9] | 86.4 [65.1 to 97.1] | 90.9 [70.8 to 98.9] | 92.1 [78.6 to 98.3] | 93.8 [69.8 to 99.8] | 100.0 [89.4 to 100.0] | 97.2 [85.5 to 99.9] | 100.0 [89.7 to 100.0] | 100.0 [78.2 to 100.0] | 92.9 [66.1 to 99.8] | 100.0 [76.8 to 100.0] | 93.3 [68.1 to 99.8] | 93.8 [69.8 to 99.8] | 92.3 [64.0 to 99.8] | 100.0 [79.4 to 100.0] | 100.0 [75.3 to 100.0] | 100.0 [78.2 to 100.0] | 100.0 [75.3 to 100.0] | 100.0 [83.2 to 100.0] | 96.0 [79.6 to 99.9]

ADVERSE EVENTS:
Time Frame: Up to 80 weeks (Parts A and B: 8 weeks or up to 16 weeks of treatment, respectively, plus 24-week follow-up; Part C: up to 16 weeks of retreatment plus 24-week follow-up)
Groups:
- A1: GT3 NC TN EBR+GZR+UPR300 (8 Wks): In Part A, participants received grazoprevir (100 mg) + uprifosbuvir (300 mg) + elbasvir (50 mg) q.d. by mouth for 8 weeks.
- A1+C: GT3 NC TN EBR+GZR+UPR300 (8 Wks); MK-3682B+RBV (16 Wks): In Part A, participants received grazoprevir (100 mg) + uprifosbuvir 300 mg) + elbasvir (50 mg) q.d. by mouth for 8 weeks. After relapsing, participants received 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d. and RBV (weight-based dosing) b.i.d. by mouth for 16 weeks in Part C.
- A2: GT3 NC TN GZR+RZR+UPR300 (8 Wks): In Part A, participants received grazoprevir (100 mg) + uprifosbuvir (300 mg) + ruzasvir (60 mg) q.d. by mouth for 8 weeks.
- A2+C: GT3 NC TN GZR+RZR+UPR300 (8 Wks); MK-3682B+RBV (16 Wks): In Part A, participants received grazoprevir (100 mg) + uprifosbuvir (300 mg) + ruzasvir (60 mg) q.d. by mouth for 8 weeks. After relapsing, participants received 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d. and RBV (weight-based dosing) b.i.d. by mouth for 16 weeks in Part C.
- A3: GT3 NC TN EBR+GZR+UPR450 (8 Wks): In Part A, participants received grazoprevir (100 mg) + uprifosbuvir (450 mg) + elbasvir (50 mg) q.d. by mouth for 8 weeks.
- A3+C: GT3 NC TN EBR+GZR+UPR450 (8 Wks); MK-3682B+RBV (16 Wks): In Part A, participants received grazoprevir (100 mg) + uprifosbuvir (450 mg) + elbasvir (50 mg) q.d. by mouth for 8 weeks. After relapsing, participants received 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d. and RBV (weight-based dosing) b.i.d. by mouth for 16 weeks in Part C.
- A4: GT3 NC TN GZR+RZR+UPR450 (8 Wks): In Part A, participants received grazoprevir 100 mg + uprifosbuvir 450 mg + ruzasvir 60 mg q.d. by mouth for 8 weeks.
- A4+C: GT3 NC TN GZR+RZR+UPR450 (8 Wks); MK-3682B+RBV (16 Wks): In Part A, participants received grazoprevir 100 mg + uprifosbuvir 450 mg + ruzasvir 60 mg q.d. by mouth for 8 weeks. After relapsing, participants received 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d. and RBV (weight-based dosing) b.i.d. by mouth for 16 weeks in Part C.
- B4: GT3 NC TN MK-3682B (8 Wks): In Part B, participants received 2 MK- 3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d. by mouth for 8 weeks.
- B5: GT3 NC TN MK-3682B + RBV (8 Wks): In Part B , participants received 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d., and RBV (weight-based dosing) b.i.d., by mouth for 8 weeks.
- B6: GT3 NC TN MK-3682B (12 Wks): In Part B, HCV GT3-infected NC TN participants received 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d. by mouth for 12 weeks.
- B7: GT3 NC TN MK-3682B + RBV (12 Wks): In Part B, HCV GT3-infected NC TN participants received 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d., and RBV (weight-based dosing) b.i.d., by mouth for 12 weeks.
- B8: GT3 NC TE MK-3682B (8 Wks): In Part B, HCV GT3-infected NC TE participants received 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d. by mouth for 8 weeks.
- B9: GT3 NC TE MK-3682B + RBV (8 Wks): In Part B, HCV GT3-infected NC TE participants received 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d., and RBV (weight-based dosing) b.i.d., by mouth for 8 weeks.
- B10: GT3 NC TE MK-3682B (12 Wks): In Part B, HCV GT3-infected NC TE participants received 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d. by mouth for 12 weeks.
- B11: GT3 NC TE MK-3682B + RBV (12 Wks): In Part B, HCV GT3-infected NC TE participants received 2 MK-3682 FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d., and RBV (weight-based dosing) b.i.d., by mouth for 12 weeks.
- B12: GT3 NC TE MK-3682B (16 Wks): In Part B, HCV GT3-infected NC TE participants received 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d. by mouth for 16 weeks.
- B13: GT3 C TN MK-3682B (12 Wks): In Part B, HCV GT3-infected C TN participants received 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d. by mouth for 12 weeks.
- B14: GT3 C TN MK-3682B + RBV (12 Wks): In Part B, HCV GT3-infected C TN participants received 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d., and RBV (weight-based dosing) b.i.d., by mouth for 12 weeks.
- B15: GT3 C TN MK-3682B (16 Wks): In Part B, HCV GT3-infected C TN participants received 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d. by mouth for 16 weeks.
- B16: GT3 C TE MK-3682B (12 Wks): In Part B, HCV GT3-infected C TE participants received 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d. by mouth for 12 weeks.
- B17: GT3 C TE MK-3682B + RBV (12 Wks): In Part B, HCV GT3-infected C TE participants received 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d., and RBV (weight-based dosing) b.i.d., by mouth for 12 weeks.
- B18: GT3 C TE MK-3682B (16 Wks): In Part B, HCV GT3-infected C TE participants received 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d. by mouth for 16 weeks.
- B19: GT3 C TE MK-3682B + RBV (16 Wks): In Part B, HCV GT3-infected C TE participants received 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d., and RBV (weight-based dosing) b.i.d., by mouth for 16 weeks.
- B20: GT4 NC TN MK-3682B (8 Wks): In Part B, HCV GT4-infected NC TN participants received 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d. by mouth for 8 weeks.
- B22: GT6 NC TN MK-3682B (12 Wks): In Part B, HCV GT6-infected NC TN participants received 2 MK-3682B FDC tablets (each containing grazoprevir 50 mg + uprifosbuvir 225 mg + ruzasvir 30 mg) q.d. by mouth for 12 weeks.
Arm/Group | A1: GT3 NC TN EBR+GZR+UPR300 (8 Wks) | A1+C: GT3 NC TN EBR+GZR+UPR300 (8 Wks); MK-3682B+RBV (16 Wks) | A2: GT3 NC TN GZR+RZR+UPR300 (8 Wks) | A2+C: GT3 NC TN GZR+RZR+UPR300 (8 Wks); MK-3682B+RBV (16 Wks) | A3: GT3 NC TN EBR+GZR+UPR450 (8 Wks) | A3+C: GT3 NC TN EBR+GZR+UPR450 (8 Wks); MK-3682B+RBV (16 Wks) | A4: GT3 NC TN GZR+RZR+UPR450 (8 Wks) | A4+C: GT3 NC TN GZR+RZR+UPR450 (8 Wks); MK-3682B+RBV (16 Wks) | B4: GT3 NC TN MK-3682B (8 Wks) | B5: GT3 NC TN MK-3682B + RBV (8 Wks) | B6: GT3 NC TN MK-3682B (12 Wks) | B7: GT3 NC TN MK-3682B + RBV (12 Wks) | B8: GT3 NC TE MK-3682B (8 Wks) | B9: GT3 NC TE MK-3682B + RBV (8 Wks) | B10: GT3 NC TE MK-3682B (12 Wks) | B11: GT3 NC TE MK-3682B + RBV (12 Wks) | B12: GT3 NC TE MK-3682B (16 Wks) | B13: GT3 C TN MK-3682B (12 Wks) | B14: GT3 C TN MK-3682B + RBV (12 Wks) | B15: GT3 C TN MK-3682B (16 Wks) | B16: GT3 C TE MK-3682B (12 Wks) | B17: GT3 C TE MK-3682B + RBV (12 Wks) | B18: GT3 C TE MK-3682B (16 Wks) | B19: GT3 C TE MK-3682B + RBV (16 Wks) | B20: GT4 NC TN MK-3682B (8 Wks) | B22: GT6 NC TN MK-3682B (12 Wks)
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/2 | 0/20 | 0/1 | 0/19 | 0/3 | 0/20 | 0/2 | 0/16 | 0/36 | 0/37 | 0/35 | 0/15 | 0/14 | 0/14 | 0/15 | 0/16 | 0/13 | 0/16 | 0/14 | 0/15 | 0/14 | 0/20 | 0/25 | 0/7 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/19 | 0/2 | 0/20 | 0/1 | 1/19 | 0/3 | 0/20 | 1/2 | 0/16 | 1/36 | 0/37 | 1/35 | 0/15 | 0/14 | 0/14 | 0/15 | 1/16 | 1/13 | 0/16 | 2/14 | 2/15 | 2/14 | 2/20 | 1/25 | 0/7 | 0/4
Other Adverse Events (participants affected / at risk) | 17/19 | 1/2 | 12/20 | 1/1 | 13/19 | 3/3 | 16/20 | 2/2 | 9/16 | 30/36 | 24/37 | 32/35 | 12/15 | 12/14 | 9/14 | 13/15 | 13/16 | 9/13 | 14/16 | 12/14 | 12/15 | 11/14 | 15/20 | 21/25 | 3/7 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A1: GT3 NC TN EBR+GZR+UPR300 (8 Wks) (N=19) | A1+C: GT3 NC TN EBR+GZR+UPR300 (8 Wks); MK-3682B+RBV (16 Wks) (N=2) | A2: GT3 NC TN GZR+RZR+UPR300 (8 Wks) (N=20) | A2+C: GT3 NC TN GZR+RZR+UPR300 (8 Wks); MK-3682B+RBV (16 Wks) (N=1) | A3: GT3 NC TN EBR+GZR+UPR450 (8 Wks) (N=19) | A3+C: GT3 NC TN EBR+GZR+UPR450 (8 Wks); MK-3682B+RBV (16 Wks) (N=3) | A4: GT3 NC TN GZR+RZR+UPR450 (8 Wks) (N=20) | A4+C: GT3 NC TN GZR+RZR+UPR450 (8 Wks); MK-3682B+RBV (16 Wks) (N=2) | B4: GT3 NC TN MK-3682B (8 Wks) (N=16) | B5: GT3 NC TN MK-3682B + RBV (8 Wks) (N=36) | B6: GT3 NC TN MK-3682B (12 Wks) (N=37) | B7: GT3 NC TN MK-3682B + RBV (12 Wks) (N=35) | B8: GT3 NC TE MK-3682B (8 Wks) (N=15) | B9: GT3 NC TE MK-3682B + RBV (8 Wks) (N=14) | B10: GT3 NC TE MK-3682B (12 Wks) (N=14) | B11: GT3 NC TE MK-3682B + RBV (12 Wks) (N=15) | B12: GT3 NC TE MK-3682B (16 Wks) (N=16) | B13: GT3 C TN MK-3682B (12 Wks) (N=13) | B14: GT3 C TN MK-3682B + RBV (12 Wks) (N=16) | B15: GT3 C TN MK-3682B (16 Wks) (N=14) | B16: GT3 C TE MK-3682B (12 Wks) (N=15) | B17: GT3 C TE MK-3682B + RBV (12 Wks) (N=14) | B18: GT3 C TE MK-3682B (16 Wks) (N=20) | B19: GT3 C TE MK-3682B + RBV (16 Wks) (N=25) | B20: GT4 NC TN MK-3682B (8 Wks) (N=7) | B22: GT6 NC TN MK-3682B (12 Wks) (N=4)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood sodium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inflammatory pseudotumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip and/or oral cavity cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A1: GT3 NC TN EBR+GZR+UPR300 (8 Wks) (N=19) | A1+C: GT3 NC TN EBR+GZR+UPR300 (8 Wks); MK-3682B+RBV (16 Wks) (N=2) | A2: GT3 NC TN GZR+RZR+UPR300 (8 Wks) (N=20) | A2+C: GT3 NC TN GZR+RZR+UPR300 (8 Wks); MK-3682B+RBV (16 Wks) (N=1) | A3: GT3 NC TN EBR+GZR+UPR450 (8 Wks) (N=19) | A3+C: GT3 NC TN EBR+GZR+UPR450 (8 Wks); MK-3682B+RBV (16 Wks) (N=3) | A4: GT3 NC TN GZR+RZR+UPR450 (8 Wks) (N=20) | A4+C: GT3 NC TN GZR+RZR+UPR450 (8 Wks); MK-3682B+RBV (16 Wks) (N=2) | B4: GT3 NC TN MK-3682B (8 Wks) (N=16) | B5: GT3 NC TN MK-3682B + RBV (8 Wks) (N=36) | B6: GT3 NC TN MK-3682B (12 Wks) (N=37) | B7: GT3 NC TN MK-3682B + RBV (12 Wks) (N=35) | B8: GT3 NC TE MK-3682B (8 Wks) (N=15) | B9: GT3 NC TE MK-3682B + RBV (8 Wks) (N=14) | B10: GT3 NC TE MK-3682B (12 Wks) (N=14) | B11: GT3 NC TE MK-3682B + RBV (12 Wks) (N=15) | B12: GT3 NC TE MK-3682B (16 Wks) (N=16) | B13: GT3 C TN MK-3682B (12 Wks) (N=13) | B14: GT3 C TN MK-3682B + RBV (12 Wks) (N=16) | B15: GT3 C TN MK-3682B (16 Wks) (N=14) | B16: GT3 C TE MK-3682B (12 Wks) (N=15) | B17: GT3 C TE MK-3682B + RBV (12 Wks) (N=14) | B18: GT3 C TE MK-3682B (16 Wks) (N=20) | B19: GT3 C TE MK-3682B + RBV (16 Wks) (N=25) | B20: GT4 NC TN MK-3682B (8 Wks) (N=7) | B22: GT6 NC TN MK-3682B (12 Wks) (N=4)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemolysis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bundle branch block right (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ocular discomfort (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pinguecula (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 2 (2) | 3 (3) | 5 (6) | 3 (4) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 1 (2) | 1 (2) | 3 (3) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Faeces soft (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infrequent bowel movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip dry (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 5 (6) | 0 (0) | 6 (6) | 0 (0) | 2 (2) | 6 (8) | 4 (5) | 5 (6) | 1 (1) | 3 (3) | 1 (1) | 2 (2) | 3 (3) | 2 (2) | 2 (3) | 3 (3) | 1 (1) | 2 (3) | 2 (2) | 4 (5) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tongue ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 2 (3) | 1 (1) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 1 (2) | 2 (2) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Energy increased (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 4 (4) | 0 (0) | 5 (5) | 0 (0) | 4 (4) | 1 (1) | 4 (4) | 1 (2) | 2 (2) | 10 (11) | 5 (5) | 13 (13) | 3 (3) | 5 (6) | 4 (4) | 5 (5) | 4 (4) | 3 (3) | 4 (5) | 3 (3) | 3 (3) | 5 (7) | 4 (4) | 9 (10) | 0 (0) | 0 (0)
Feeling abnormal (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling jittery (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Local swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Vessel puncture site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Genital herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infected dermal cyst (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periodontitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (2) | 2 (3) | 0 (0) | 2 (2) | 6 (7) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 3 (3) | 4 (4) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Wound infection staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 8 (8) | 1 (1) | 5 (5) | 1 (1) | 6 (6) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foreign body (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial test positive (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood potassium increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Protein urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cells urine positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperlipasaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyskinesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 4 (5) | 1 (3) | 5 (6) | 1 (2) | 5 (8) | 0 (0) | 5 (6) | 1 (1) | 5 (6) | 12 (13) | 7 (7) | 8 (8) | 2 (2) | 5 (5) | 2 (2) | 5 (6) | 6 (6) | 1 (1) | 4 (4) | 4 (5) | 1 (1) | 2 (3) | 3 (3) | 9 (11) | 1 (1) | 2 (2)
Hypersomnia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Parosmia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Poor quality sleep (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tension headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Affect lability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Emotional disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (3) | 0 (0) | 1 (2) | 1 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Tearfulness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal cyst (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast tenderness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulval haematoma (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 2 (2) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 4 (5) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Macule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 5 (5) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 1 (3) | 1 (1) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arteriosclerosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation.